CLINICAL TRIAL: NCT02271477
Title: Can Vena Cava Ultrasound Guided Volume Repletion Prevent Spinal Induced Significant Hypotension in Elective Surgical Patients? A Randomized, Case Control, Prospective Trial.
Brief Title: Can Vena Cava Ultrasound Guided Volume Repletion Prevent Spinal Induced Significant Hypotension in Elective Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CERU-1402
Record Dates: First submitted 2014-10-10; First posted 2014-10-22 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2015-04

CONDITIONS: Fluid Overload; Anesthesia; Adverse Effect, Spinal and Epidural; Regional Anesthesia Morbidity
Keywords: Fluid replacement; Trans-Thoracic Echocardiography; Spinal Anesthesia; Empirical Volemic Repletion
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wild-Type (No Intervention): The setting is standard spinal anesthesia and corresponds to our first arm of the study, used as the control sample and statistical reference. During the induction phase, the patient is fitted with non-invasive blood pressure monitoring, three-lead ECG, pulse-oximetry and peripheral intravenous device. Data and vital signs are recorded and an infusion of crystalloid (NaCl 0.9% or Ringer's acetate) is given during the procedure until the beginning of the operation. Total amount of fluid is also recorded before and after the spinal anesthesia.
- Echocardiography (Experimental): In addition to the current clinical standard, a Trans-Thoracic Echocardiography is performed before spinal anesthesia, with the aim of assessing the patient's volume status; the exam is performed to assess size and collapsing of the Inferior Vena Cava during breathing cycle. According to different pre-established parameters13, the patient is defined as fluid-responsive or unresponsive. If the patient is not responsive, investigators proceed to spinal anesthesia; otherwise they proceed to administration of crystalloid bolus (500 ml of NaCl 0.9% or Hartmann's solution). The patient may receive another bolus so as to reach a non-responsive pattern for echocardiographic evaluation.
  Interventions: Device: Ultrasound-guided volemic repletion

INTERVENTIONS:
Device: Ultrasound-guided volemic repletion — After echocardiography analysis of Inferior Vena Cava, patient is repleted with a pre-established bolus of fluid (500 ml of crystalloid). After this repletion, patient is analyzed till the exam reach signal of non-responsiveness, previously defined as a reduction of Inferior Vena Cava diameter less than 36% from baseline level during normal breath
  Other Names: IVCUS
  Arms: Echocardiography

SUMMARY:
Aim of this study is to determine whether Inferior Vena Cava analyzed by trans-thoracic echocardiography is an effective method to guide titrated fluid repletion in non critical patients, in order both to decrease post procedural significant hypotension rate and to avoid unnecessary fluid overload in patients undergoing spinal anesthesia for elective surgical procedures

DETAILED DESCRIPTION:
The setting is standard spinal anesthesia and corresponds to our first arm of the study, used as the control sample and statistical reference. During the induction phase, the patient is fitted with non-invasive blood pressure monitoring, three-lead ECG, pulse-oximetry and peripheral intravenous device. Data and vital signs are recorded and an infusion of crystalloid (NaCl 0.9% or Ringer's acetate) is given during the procedure until the beginning of the operation. Total amount of fluid is also recorded before and after the spinal anesthesia.

In addition to the current clinical standard, for the second arm of the study, a trans-thoracic echocardiography is performed before spinal anesthesia, with the aim of assessing the patient's volume status; the exam is performed to assess size and collapsing of the Inferior Vena Cava during breathing cycle. According to different pre-established parameters, the patient is defined as fluid-responsive or unresponsive. If the patient is not responsive, investigators proceed to spinal anesthesia; otherwise they proceed to administration of crystalloid bolus (500 ml of NaCl 0.9% or Hartmann's solution). The patient may receive another bolus so as to reach a non-responsive pattern for echocardiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* grater than 18 year old
* requiring spinal anesthesia
* classified according to American Society of Anesthesiology (ASA) level as 1, 2 or 3

Exclusion Criteria:

* patients required invasive blood pressure monitoring (arterial/pulmonary catheter, thermodilution catheter),
* patients show signs of pre-procedural hypotension (defined as two measurements of systolic arterial pressure less than 80 mmHg and/or mean arterial pressure less than 60 mmHg),
* patients unable to give informed consent to language barriers, mental retard or any reduction in own ability to understand or give their informed consent,
* patient in which is not possible to perform spinal anesthesia for patient's refusal or technical difficulties in sampling,
* patients with International Normalized Ratio (INR) greater than 1.5 and/or activated Partial Thrombin Time in therapeutic range (more than 1.5 - 2 times the patient's normal values) and/or anti-factor X activity in therapeutic range
* patients with thrombocytopenia less than 50 G/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuele Ceruti, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Ospedale Regionale di Bellinzona e Valli (ORBV) - Sede Bellinzona, Bellinzona, Switzerland

REFERENCES:
- [Result] Antonelli M, Levy M, Andrews PJ, Chastre J, Hudson LD, Manthous C, Meduri GU, Moreno RP, Putensen C, Stewart T, Torres A. Hemodynamic monitoring in shock and implications for management. International Consensus Conference, Paris, France, 27-28 April 2006. Intensive Care Med. 2007 Apr;33(4):575-90. doi: 10.1007/s00134-007-0531-4. PMID 17285286
- [Result] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Result] Kim HJ, Kim JS. A cardiovascular collapse following vigorous cough during spinal anesthesia. Korean J Anesthesiol. 2013 Dec;65(6 Suppl):S49-50. doi: 10.4097/kjae.2013.65.6S.S49. No abstract available. PMID 24478870
- [Result] Nogueira CS, Lima LC, Paris VC, Neiva PM, Otani ET, Couceiro Rde O, Burim F, Ferreira JA Jr, Cadecaro P. A comparative study between bupivacaine (S75-R25) and ropivacaine in spinal anesthesia for labor analgesia. Rev Bras Anestesiol. 2010 Sep-Oct;60(5):484-94. doi: 10.1016/S0034-7094(10)70060-X. English, Portuguese. PMID 20863929
- [Result] Cherpanath TG, Geerts BF, Lagrand WK, Schultz MJ, Groeneveld AB. Basic concepts of fluid responsiveness. Neth Heart J. 2013 Dec;21(12):530-6. doi: 10.1007/s12471-013-0487-7. PMID 24170232
- [Result] Jabalameli M, Soltani HA, Hashemi J, Behdad S, Soleimani B. Prevention of post-spinal hypotension using crystalloid, colloid and ephedrine with three different combinations: A double blind randomized study. Adv Biomed Res. 2012;1:36. doi: 10.4103/2277-9175.100129. Epub 2012 Aug 28. PMID 23326767
- [Result] Xu S, Wu H, Zhao Q, Shen X, Guo X, Wang F. The median effective volume of crystalloid in preventing hypotension in patients undergoing cesarean delivery with spinal anesthesia. Rev Bras Anestesiol. 2012 May-Jun;62(3):312-24. doi: 10.1016/S0034-7094(12)70132-0. PMID 22656677
- [Result] Buggy DJ, Power CK, Meeke R, O'Callaghan S, Moran C, O'Brien GT. Prevention of spinal anaesthesia-induced hypotension in the elderly: i.m. methoxamine or combined hetastarch and crystalloid. Br J Anaesth. 1998 Feb;80(2):199-203. doi: 10.1093/bja/80.2.199. PMID 9602585
- [Result] Vieillard-Baron A, Chergui K, Rabiller A, Peyrouset O, Page B, Beauchet A, Jardin F. Superior vena caval collapsibility as a gauge of volume status in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1734-9. doi: 10.1007/s00134-004-2361-y. Epub 2004 Jun 26. PMID 15375649
- [Result] Zollei E, Bertalan V, Nemeth A, Csabi P, Laszlo I, Kaszaki J, Rudas L. Non-invasive detection of hypovolemia or fluid responsiveness in spontaneously breathing subjects. BMC Anesthesiol. 2013 Nov 5;13(1):40. doi: 10.1186/1471-2253-13-40. PMID 24188480
- [Result] Barbier C, Loubieres Y, Schmit C, Hayon J, Ricome JL, Jardin F, Vieillard-Baron A. Respiratory changes in inferior vena cava diameter are helpful in predicting fluid responsiveness in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1740-6. doi: 10.1007/s00134-004-2259-8. Epub 2004 Mar 18. PMID 15034650
- [Result] Zhang Z, Xu X, Ye S, Xu L. Ultrasonographic measurement of the respiratory variation in the inferior vena cava diameter is predictive of fluid responsiveness in critically ill patients: systematic review and meta-analysis. Ultrasound Med Biol. 2014 May;40(5):845-53. doi: 10.1016/j.ultrasmedbio.2013.12.010. Epub 2014 Feb 2. PMID 24495437
- [Result] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199
- [Result] Muller L, Bobbia X, Toumi M, Louart G, Molinari N, Ragonnet B, Quintard H, Leone M, Zoric L, Lefrant JY; AzuRea group. Respiratory variations of inferior vena cava diameter to predict fluid responsiveness in spontaneously breathing patients with acute circulatory failure: need for a cautious use. Crit Care. 2012 Oct 8;16(5):R188. doi: 10.1186/cc11672. PMID 23043910
- [Result] Chinachoti T, Tritrakarn T. Prospective study of hypotension and bradycardia during spinal anesthesia with bupivacaine: incidence and risk factors, part two. J Med Assoc Thai. 2007 Mar;90(3):492-501. PMID 17427526
- [Result] Slama M, Masson H, Teboul JL, Arnout ML, Susic D, Frohlich E, Andrejak M. Respiratory variations of aortic VTI: a new index of hypovolemia and fluid responsiveness. Am J Physiol Heart Circ Physiol. 2002 Oct;283(4):H1729-33. doi: 10.1152/ajpheart.00308.2002. Epub 2002 Jun 20. PMID 12234829
- [Derived] Ceruti S, Anselmi L, Minotti B, Franceschini D, Aguirre J, Borgeat A, Saporito A. Prevention of arterial hypotension after spinal anaesthesia using vena cava ultrasound to guide fluid management. Br J Anaesth. 2018 Jan;120(1):101-108. doi: 10.1016/j.bja.2017.08.001. Epub 2017 Nov 23. PMID 29397116

RESULTS

PARTICIPANT FLOW:
Groups:
- Echocardiography: In addition to the current clinical standard, a Trans-Thoracic Echocardiography is performed before spinal anesthesia, with the aim of assessing the patient's volume status; the exam is performed to assess size and collapsing of the Inferior Vena Cava during breathing cycle. According to different pre-established parameters13, the patient is defined as fluid-responsive or unresponsive. If the patient is not responsive, investigators proceed to spinal anesthesia; otherwise they proceed to administration of crystalloid bolus (500 ml of NaCl 0.9% or Hartmann's solution). The patient may receive another bolus so as to reach a non-responsive pattern for echocardiographic evaluation.
  After echocardiography analysis of Inferior Vena Cava, patient is repleted with a pre-established bolus of fluid (500 ml of crystalloid). After this repletion, patient is analyzed till the exam reach signal of non-responsiveness, previously defined as a reduction of Inferior Vena Cava diameter less than 36%
Period: Overall Study
Arm/Group | Wild-Type | Echocardiography
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Echocardiography: In addition to the current clinical standard, a Trans-Thoracic Echocardiography is performed before spinal anesthesia, with the aim of assessing the patient's volume status; the exam is performed to assess size and collapsing of the Inferior Vena Cava during breathing cycle. According to different pre-established parameters13, the patient is defined as fluid-responsive or unresponsive. If the patient is not responsive, investigators proceed to spinal anesthesia; otherwise they proceed to administration of crystalloid bolus (500 ml of NaCl 0.9% or Hartmann's solution). The patient may receive another bolus so as to reach a non-responsive pattern for echocardiographic evaluation. After echocardiography analysis of Inferior Vena Cava, patient is repleted with a pre-established bolus of fluid (500 ml of crystalloid).
- Total: Total of all reporting groups
Arm/Group | Wild-Type | Echocardiography | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (16.7) | 56.6 (18.8) | 57.74 (18.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 36 | 37 | 73
Weight [Mean (Standard Deviation); unit: Kg] | 78.01 (18.40) | 76.07 (17.59) | 76.52 (25)
Systolic blood pressure (SBP) pre-induction [Mean (Standard Deviation); unit: mmHg] — This is the blood pressure recorder at the entrance in the operative block. The measure is the international unit of measure: mmHg
  mmHg | 136 (22) | 132 (21) | 134.05 (21.95)
Mean blood pressure (MBP) pre-induction [Mean (Standard Deviation); unit: mmHg] — This is the mean blood pressure recorder at the entrance in the operative block. The measure is the international unit of measure: mmHg
  mmHg | 94.5 (13.99) | 91.5 (13) | 93 (13.21)
Heart Rate (HR) pre-induction [Mean (Standard Deviation); unit: bpm] | 70 (16) | 72 (12) | 71.88 (12.27)
B-blockers therapy [Number; unit: participants] — Chronic assumption of B-blockers therapy prior to the procedure
  participants
    B-blockers | 7 | 1 | 8
    No therapy | 73 | 79 | 152
ACE-inhibitors therapy [Number; unit: participants] — Chronic assumption of ACE-inhibitors therapy prior to intervention
  participants
    ACE-inhibitors | 9 | 5 | 14
    No therapy | 71 | 75 | 146
Crystalloid therapy [Number; unit: participants] — Use of crystalloid therapy during the procedure
  participants | 80 | 80 | 160
Type of crystalloid therapy [Number; unit: participants] — Type of crystalloid used during the procedure
  participants
    Ringer | 80 | 80 | 160
    NaCl 0.9% | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Arterial Hypotension
Description: To compare rates of arterial hypotension (previously define by international standard) after spinal anesthesia in patients who have undergone volemic optimization according to Trans-thoracic Echocardiography with patients who have been treated according to the current standard on the intention to treat population.
Time Frame: 30 minute after spinal anesthesia
Population: Rate of arterial hypotension after standardized spinal anesthesia
Measure: Number; unit: percentage of participants
Arm/Group | Wild-Type | Echocardiography
Number analyzed (Participants) | 80 | 80
percentage of participants | 42.5 | 27.5

2. Secondary Outcome: Total Amount of IV Fluid at the End of the Procedure
Description: To assess if there is a difference between all treatments in the total quantity of fluids amount
Time Frame: 30 minutes after spinal anesthesia
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Groups:
- Echocardiography: In addition to the current clinical standard, a Trans-Thoracic Echocardiography is performed before spinal anesthesia, with the aim of assessing the patient's volume status; the exam is performed to assess size and collapsing of the Inferior Vena Cava during breathing cycle. According to different pre-established parameters13, the patient is defined as fluid-responsive or unresponsive. If the patient is not responsive, investigators proceed to spinal anesthesia; otherwise they proceed to administration of crystalloid bolus (500 ml of NaCl 0.9% or Hartmann's solution). The patient may receive another bolus so as to reach a non-responsive pattern for echocardiographic evaluation.
  Ultrasound-guided volemic repletion: After echocardiography analysis of Inferior Vena Cava, patient is repleted with a pre-established bolus of fluid (500 ml of crystalloid). After this repletion, patient is analyzed till the exam reach signal of non-responsiveness
Arm/Group | Wild-Type | Echocardiography
Number analyzed (Participants) | 80 | 80
milliliters (mL) | 350 [200 to 550] | 665 [250 to 800]

3. Secondary Outcome: Percentage of Participants Administered Vasoactive Drug
Description: Total amount of vasoactive drug administered for each group; for "vasoactive drug" we intended the use both of atropine than vascular amine
Time Frame: 30 minutes after spinal anesthesia
Measure: Number; unit: percentage of participants
Arm/Group | Wild-Type | Echocardiography
Number analyzed (Participants) | 80 | 80
percentage of participants | 13.51 | 6.49

4. Secondary Outcome: Time of Procedures
Description: Time employed to execute all procedure from the start of the study till 30 minutes after the end of the procedure
Time Frame: From time 0 to 30 minutes after spinal anesthesia
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wild-Type | Echocardiography
Number analyzed (Participants) | 80 | 80
minutes | 22 (13) | 24 (10)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events are checked till the end of the surgical procedure.
Description: Serious Adverse Events are defined as all possible complication related to hypotension after spinal anaesthesia (neurological deficit related to hypotension, chest pain, myocardial ischemia/infarction, renal failure, cardiac arrest) is checked till the end of the surgical procedure.
Groups:
- Echocardiography: In addition to the current clinical standard, a Trans-Thoracic Echocardiography is performed before spinal anesthesia, with the aim of assessing the patient's volume status; the exam is performed to assess size and collapsing of the Inferior Vena Cava during breathing cycle. According to different pre-established parameters13, the patient is defined as fluid-responsive or unresponsive. If the patient is not responsive, investigators proceed to spinal anesthesia; otherwise they proceed to administration of crystalloid bolus (500 ml of NaCl 0.9% or Hartmann's solution). The patient may receive another bolus so as to reach a non-responsive pattern for echocardiographic evaluation. Ultrasound-guided volemic repletion: After echocardiography analysis of Inferior Vena Cava, patient is repleted with a pre-established bolus of fluid (500 ml of crystalloid).
Arm/Group | Wild-Type | Echocardiography
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

LIMITATIONS AND CAVEATS:
It cannot be performed blindly. Ultrasound is an operator-dependent technique.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes